CLINICAL TRIAL: NCT03350113
Title: Integration of Clinical and Laboratory Information to Generate Technological Advance for the Diagnosis of Sepsis - The Intelligence 2 Trial
Brief Title: Hemospec Device for Sepsis Diagnosis
Acronym: INTELLIGENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Collaborators: General Hospital of Lamia (Other); University of Jena (Other)
Responsible Party: Principal Investigator, Evangelos J. Giamarellos-Bourboulis, M.D., Associate Professor of Internal Medicine, University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INTELLIGENCE2
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Sepsis
Keywords: prognosis; diagnosis
MeSH Terms: conditions — Sepsis; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HemoSpec (Experimental): Blood Sampling for analysis in the HemoSpec device
  Interventions: Device: Blood sampling for analysis

INTERVENTIONS:
Device: Blood sampling for analysis — Blood Sampling for Analysis
  Other Names: Hemospec

SUMMARY:
A diagnostic devise, namely HemoSpec, had been developed that integrates clinical information, along with information on circulating protein biomarkers and the morphology of white blood cells to achieve early diagnosis of sepsis. The current study is aiming to validate and improve performance of HemoSpec for the rapid assessment of the critically ill patient in the Emergency Department.

DETAILED DESCRIPTION:
Sepsis is a life-threating organ dysfunction resulting from the dysregulated response of the host to an infection. It is estimated that 1.5 million people present with sepsis annually in Northern America and another 1.5 million people in Europe; 30 to 50% of them die making sepsis the leading cause of death. The key-point in the management of sepsis is the early resuscitation with broad- spectrum antimicrobials and intravenous fluids, if possible within the first hour. However, it is not easy to achieve this goal, especially among patients assessed in the Emergency Department (ED), as the diagnosis of an infection is often delayed until the patient's laboratory and imaging tests are completed.

In an attempt to improve the failure of physicians for early sepsis recognition in the ED, several markers have been developed. The most widely used biomarkers are the absolute number of neutrophils, C-reactive protein (CRP) and procalcitonin (PCT). HemoSpec is a device capable of incorporating clinical information from the patient with laboratory data. The analysis provides information on white blood cell morphology, CRP, PCT, interleukin (IL) -6 and suPAR. The device software has been created from all of the above information collected from prospective cohorts of patients from Greece and Germany. The diagnostic function of HemoSpec has so far been validated in two Phase II studies. The first study took place in Germany and involved 60 patients (20 controls, 20 with systemic inflammatory response and 20 with sepsis) who were hospitalized at the University Hospital in Jena. The second study is currently being conducted in Greece and aims to use the information from the HemoSpec device for the prospective categorization of patients with confirmed infection in patients with sepsis and in patients without sepsis.

The above two studies share a common Phase II design in order to validate HemoSpec's diagnostic ability among patients who are clinically diagnosed with sepsis. The clinical reliability of HemoSpec can be verified in a multicenter prospective trial involving patients assessed in the ED. The present study aims to assess the diagnostic ability of the device in ED patients with clinical signs of infection who have a significant risk of death that makes them likely to suffer from sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Admission in the Emergency Department
* Age above or equal to 18 years old
* Both genders
* Written consent provided from patients or their first-degree relatives for patients unable to consent
* Considerable risk of death as indicated by the presence of at least one of the following: i) sudden alteration of mental status; ii) systolic blood pressure less than 100 mmHg; and iii) high respiratory rate defined as more than or equal to 22 breaths per minute.

Exclusion Criteria:

* Known infection by the human immunodeficiency virus-1
* Acute myocardial infarction as evidenced by the electrocardiographic finding of ST- elevation.
* Single trauma or multiple injuries
* Known pregnancy and breastfeeding
* Patients with a life expectancy of less than 28 days and with limited treatment options

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity of HemoSpec for the diagnosis of sepsis | 4 days
  The sensitivity of HemoSpec output to diagnose the presence of sepsis compared to the absence of sepsis. HemoSpec output will be considered to provide a satisfactory diagnosis of sepsis if sensitivity for the diagnosis is greater than 90%.

SECONDARY OUTCOMES:
Diagnostic performance for sepsis | 4 days
  The diagnostic performance of HemoSpec output to diagnose the presence of sepsis compared to the absence of sepsis. The diagnostic performance is composed by the aggregation of specificity, positive predictive value and negative predictive value.
Prognostics performance for sepsis | 28 days
  The prognostic performance of HemoSpec output to predict unfavorable outcome compared to survivors. The prognostic performance is composed by the aggregation of sensitivity, specificity, positive predictive value and negative predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos J Giamarellos-Bourboulis, MD, PhD, Study Chair — National and Kapodistrian University of Athens; Magdalini Bristianou, MD, PhD, Principal Investigator — General Hospital of Lamia; Michael Bauer, MD, PhD, Principal Investigator — Jena University Hospital
Locations (3):
- Univeristy of Jena, Jena, Germany
- Greece (2):
  - General Hospital of Lamia, Lamia, Phthiotis
  - 4th Department of Internal Medicine, ATTIKON University Hospital, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Becker KL, Snider R, Nylen ES. Procalcitonin assay in systemic inflammation, infection, and sepsis: clinical utility and limitations. Crit Care Med. 2008 Mar;36(3):941-52. doi: 10.1097/CCM.0B013E318165BABB. PMID 18431284
- [Result] Giamarellos-Bourboulis EJ, Norrby-Teglund A, Mylona V, Savva A, Tsangaris I, Dimopoulou I, Mouktaroudi M, Raftogiannis M, Georgitsi M, Linner A, Adamis G, Antonopoulou A, Apostolidou E, Chrisofos M, Katsenos C, Koutelidakis I, Kotzampassi K, Koratzanis G, Koupetori M, Kritselis I, Lymberopoulou K, Mandragos K, Marioli A, Sunden-Cullberg J, Mega A, Prekates A, Routsi C, Gogos C, Treutiger CJ, Armaganidis A, Dimopoulos G. Risk assessment in sepsis: a new prognostication rule by APACHE II score and serum soluble urokinase plasminogen activator receptor. Crit Care. 2012 Aug 8;16(4):R149. doi: 10.1186/cc11463. PMID 22873681